CLINICAL TRIAL: NCT04845503
Title: Stereotactic MRI-guided Radiation Therapy for Localized prostatE Cancer
Acronym: SMILE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Heidelberg (Other)
Collaborators: Ludwig-Maximilians - University of Munich (Other); University Hospital, Zürich (Other)
Responsible Party: Principal Investigator, Juergen Debus, Medical Director RadioOncology, University Hospital Heidelberg
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SMILE
Record Dates: First submitted 2021-03-05; First posted 2021-04-15 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- MR-guided Radiotherapy (5 x 7,5 Gy) (Experimental): 5 x 7,5 Gy prescribed on the PTV
  Interventions: Radiation: MR-guided Radiotherapy

INTERVENTIONS:
Radiation: MR-guided Radiotherapy — Total Dose 37,5 Gy, Single Dose 7,5 Gy, 5 Fractions applied in 1-2 weeks

SUMMARY:
As the most common carcinoma in men, prostate cancer is a significant tumor entity in oncology. In addition to the surgical approach, definitive radiotherapy is an equivalent therapy alternative in the non-metastatic primary situation. However, radiotherapy usually stretches over a period of several weeks (7 to 8 weeks) during which the patient receives irradiation on a daily basis. For this reason and for radiobiological considerations the total treatment time is increasingly shortened. It has been shown in several randomized phase III studies that shorting radiotherapy to about 4 weeks by increasing the single dose (so-called hypofractionation) is possible. Meanwhile there is also more data on extreme hypofractionation (max. 10 radiation sessions) available, however often times, extensive preparations are necessary (such as the invasive introduction of markers into the prostate). The current, prospective, non-randomized, multicentric, Phase II SMILE study is now testing whether the MRI-guided radiotherapy with a greatly shortened radiotherapy of the prostate over 5 radiation sessions is possible and safe.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed prostate carcinoma with tissue classification according to Gleason score and PSA
* low- or intermediate-risk carcinoma according to d'Amico criteria or early high-risk Carcinoma (cT3a and / or GS ≤ 8 and / or PSA ≤ 20ng / ml)
* IPSS (International Prostate Symptom Score) max. 12
* Prostate volume <80cm³
* Karnofsky index ≥ 70%
* Age ≥ 18 years
* Patient information provided and written consent
* Ability of the patient to give consent

Exclusion Criteria:

* Previous radiotherapy in the pelvis
* Previous local therapy of the prostate
* lymphogenic metastasis
* Stage IV (distant metastases)
* Contraindication to MRI
* Simultaneous participation in another clinical study which could influence results of either of the respective study

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2021-03-25 (Actual); Primary Completion 2023-03-25 (Actual); Study Completion 2028-03-25 (Estimated)

PRIMARY OUTCOMES:
Toxicity or Discontinuation of Therapy | Within 1 Year
  One of the the following events are counted as an Event (Number of Participants affected):
  * any urogenital or gastrointestinal grade ≥ 2 toxicity within one year after the start of RT (according to NCI CTCAE Version 5.0)
  * Discontinuation of therapy, with a connection to the study treatment

SECONDARY OUTCOMES:
Mortality | Within 1 year and within 5 years
  Mortality due to study treatment or due to prostate Cancer (Number of Participants deceased)
Number of Toxicities | Within 1 year and within 5 years after start of radiotherapy
  Number and severity of urogenital or gastrointestinal toxicity
bPFS | from start of radiotherapy (day 1) until PSA-relapse according to Phoenix-Criteria (Prostate-specific antigen (PSA) nadir + 2 ng/mL after radiotherapy), assessed up to 5 years
  biochemical progression free survival
Hormone therapy-free Survival | from start of radiotherapy until start of hormon treatment; maximum 3 months neoadjuvant
  Hormone therapy-free Survival
OS | from start of radiotherapy (day 1) until death or censoring assessed up to 5 years
  overall survival
Quality of life according to EORTC QLQ-C30 | from start of radiotherapy (day 1) until end of follow-up (up to 5 years)
  Quality of life according to EORTC QLQ-C30
Quality of life according to EORTC QLQ-PR25 | from start of radiotherapy (day 1) until end of follow-up (up to 5 years)
  Quality of life according to EORTC QLQ-PR25
Symptoms and Toxicity | from start of radiotherapy (day 1) until end of follow-up (up to 5 years)
  Symptoms and Toxicity according to NCI CTCAE (Rate)

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Heidelberg, Radiation Oncology, Heidelberg, Germany

IPD SHARING:
Plan to Share IPD: No